CLINICAL TRIAL: NCT01939288
Title: Effect of Neuromuscular Calf Stimulation and Intermittent Pneumatic Compression on Lower Limb Venous Hemodynamics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: JROHH0324
Record Dates: First submitted 2013-08-08; First posted 2013-09-11 (Estimated); Results first posted 2019-07-22 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Intermittent Pneumatic Compression
Keywords: neuromuscular stimulation; intermittent pneumatic compression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Half of recruited subjects (n=5)
  Interventions: Device: Neuromuscular stimulation, followed by intermittent pneumatic compression
- Group 2 (Experimental): Other half of recruited subjects (n=5)
  Interventions: Device: Intermittent pneumatic compression, followed by neuromuscular stimulation

INTERVENTIONS:
Device: Neuromuscular stimulation, followed by intermittent pneumatic compression
  Other Names: Device 1 followed by a break, followed by device 2
  Arms: Group 1
Device: Intermittent pneumatic compression, followed by neuromuscular stimulation
  Other Names: Device 2, followed by a short break then device 2
  Arms: Group 2

SUMMARY:
What is known?

* Disorders of peripheral circulation result in vascular morbidity and mortality
* Augmentation of peripheral circulation has been shown to be of benefit in both venous and arterial disease
* The benefit of intermittent pneumatic compression is clinically well evidenced.
* The use of intermittent pneumatic compression is limited by compliance issues related to sleeve application and external power source.

What new information will this trial contribute?

- This evaluates the haemodynamic effect of a new electrical device for augmentation of peripheral circulation

DETAILED DESCRIPTION:
RATIONALE - Enhancement of peripheral circulation has been shown to be of benefit in many vascular disorders, and the clinical effectiveness of intermittent pneumatic compression (IPC) is well established in peripheral vascular disease.

OBJECTIVE - This study aims to compare the haemodynamic efficacy of a novel neuromuscular electrical stimulation (NMES) device with IPC in healthy subjects.

METHODS - 10 healthy volunteers will be randomised into two groups, in an interventional cross-over trial. Baseline measurements of haemodynamic velocity and flow will be taken, then subjects given bilateral therapy with each of the two devices in turn. Laser doppler fluximetry readings will be taken from the hand and foot. Baseline readings will be compared with readings taken after immediate cessation of therapy, and after 10 minutes. Tolerability will be measured using a verbal reported score.

ELIGIBILITY:
Inclusion Criteria

Age >18 yrs, Body Mass Index (BMI) 17-30Kg/m2

Exclusion Criteria

History of heart disease or respiratory disorder, pregnancy, history of peripheral vascular disease or previous thromboembolic event, ABPI< 0.9, cardiac pacemaker, history of leg fractures and/or presence of metal implants in the leg, long distance travel within one week prior to study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kate Williams, Principal Investigator — Imperial College London
Locations (1):
- Academic Vascular Surgery, Charing Cross Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Williams KJ, Moore HM, Davies AH. Haemodynamic changes with the use of neuromuscular electrical stimulation compared to intermittent pneumatic compression. Phlebology. 2015 Jun;30(5):365-72. doi: 10.1177/0268355514531255. Epub 2014 Apr 10. PMID 24722790
- See also: PI information — http://www.imperial.ac.uk/people/k.williams

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Half of recruited subjects (n=5)
  Neuromuscular stimulator followed by IPC
- Group 2: Other half of recruited subjects (n=5)
  IPC followed by neuromuscular stimulator
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Healthy
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.1 (3.8) | 27.1 (3.8) | 27.1 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: IPC(on) Peak Velocity Change From Baseline
Description: Ultrasound measurements of peak velocity. This is taken from the left leg superficial femoral vein and artery
Time Frame: One day
Measure: Median (Inter-Quartile Range); unit: cm/s
Groups:
- Overall Summation: Grouping all subject together so that no one intervention in a certain order skews results
Arm/Group | Overall Summation
Number analyzed (Participants) | 10
cm/s | 6.2 [0.1 to 16.5]

2. Other Pre Specified Outcome: NMES(on) Peak Velocity Change From Baseline
Time Frame: One day
Measure: Median (Inter-Quartile Range); unit: cm/s
Arm/Group | Overall Summation
Number analyzed (Participants) | 10
cm/s | 36.7 [18.8 to 49.1]

ADVERSE EVENTS:
Time Frame: 10 days
Groups:
- Group 1: Neuromuscular stimulator
- Group 2: Intermittent pneumatic compression
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes